CLINICAL TRIAL: NCT00908505
Title: Comparison Between bi-Phasic Negative Pressure Ventilator Therapy and Physiotherapy in Cystic Fibrosis Patients
Brief Title: Comparison Between RTX (Biphasic Cuirass Ventilator) and Physiotherapy in Cystic Fibrosis Patients
Acronym: RTX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Arik Tzukert, DMD, Hadassah Medical Organization, Jerusalem, Israel
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RTX- HMO-CTIL
Record Dates: First submitted 2009-05-19; First posted 2009-05-27 (Estimated); Last update posted 2009-05-27 (Estimated); Status verified 2009-05

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; physiotherapy; pulmonary function test
MeSH Terms: conditions — Cystic Fibrosis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- physiotherapy (Experimental)
  Interventions: Procedure: physiotherapy

INTERVENTIONS:
Procedure: physiotherapy — physiotherapy either by biphasic cuirass ventilator or physiotherapist

SUMMARY:
The purpose of this study is to compare the effectiveness of different mucous clearance techniques in cystic fibrosis patients

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is associated with chronic progressive lung disease that may lead to respiratory failure.Bi-Phasic Cuirass Ventilation (BPCV) is a form of non-invasive respiratory support, which can provide negative pressure ventilation as well as high frequency chest wall oscillations and cough mode.The standard therapy for CF patients to release mucous is treatment by a physiotherapist. In this study we will compare the effect of BPCV with regular physiotherapy by full pulmonary function testing prior and post treatment.

ELIGIBILITY:
Inclusion Criteria:

* CF patients over 7 years old

Exclusion Criteria:

* Hemoptysis
* Pregnancy

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function test | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: David Shoseyov, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel